CLINICAL TRIAL: NCT00458731
Title: Phase I Clinical Trial Evaluating the Toxicity, Pharmacokinetics and Biological Effect of Intravenous Bevacizumab (Avastin TM) in Combination With Escalating Doses of Oral AZD2171 for Patients With Advanced Malignancies
Brief Title: Bevacizumab and Cediranib Maleate in Treating Patients With Metastatic or Unresectable Solid Tumor, Lymphoma, Intracranial Glioblastoma, Gliosarcoma or Anaplastic Astrocytoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00184; NCI-2009-00184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MDACC 2005-0910; CDR0000538277; MDACC 2005-0910 (Other: M D Anderson Cancer Center); 7534 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2013-12

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Progressive Hairy Cell Leukemia, Initial Treatment; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Hodgkin Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Recurrence; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Bevacizumab; cediranib

ARMS (1):
- Treatment (cediranib maleate and bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral cediranib maleate once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of bevacizumab and cediranib maleate until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Biological: bevacizumab; Drug: cediranib maleate

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin

SUMMARY:
This phase I trial is studying the side effects and best dose of bevacizumab and cediranib maleate in treating patients with metastatic or unresectable solid tumor, lymphoma, intracranial glioblastoma, gliosarcoma or anaplastic astrocytoma. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Cediranib maleate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Bevacizumab and cediranib maleate may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving bevacizumab together with cediranib maleate may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity profile of intravenous bevacizumab (avastin) administered in combination with oral AZD2171 (cediranib maleate) for patients with advanced malignancies.

II. To determine the pharmacokinetic profile of oral AZD2171 in combination with bevacizumab (avastin) administered to patients with advanced malignancies.

SECONDARY OBJECTIVES:

I. To evaluate the serum concentrations of Nitric Oxide (NO) and Nitric oxide synthase (NOS) among patients treated with this regimen and to correlate with VEGF expression.

II. To determine changes in the tumor vasculature detected by DCE-MRI among patients treated with this combination of VEGF receptor blocking agents.

III. To evaluate the potential predictive role of angiogenesis molecular endpoints in malignant effusion samples.

IV. To assess in a descriptive fashion the efficacy of the studied regimen.

OUTLINE: This is a dose-escalation study.

Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral cediranib maleate once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bevacizumab and cediranib maleate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Blood samples are acquired at baseline, on day 2, and after 2 courses of treatment for pharmacokinetic studies. Samples are analyzed by TUNEL, immunofluorescence staining, laser-scanning cytometry, flow cytometry, enzyme-linked immunosorbent assay, and immunohistochemistry to assess apoptosis in tumor and endothelial cells, microvessel density mean vessel volume, nitric oxide concentration, and signal transduction pathways (i.e., ERK ½, P38 mitogen-activated protein kinase, protein kinase B, circulating endothelial and progenitor cells, basic fibroblast growth factor, vascular endothelial growth factor (VEGF) receptor phosphorylation, VEGF, and hypoxia inducible factor-1α). Some patients also undergo tissue biopsy at baseline and after 2 courses of treatment for characterization of vascular and angiogenesis markers. Some patients also undergo DCE-MRI at baseline, once between days 22-24, and after every 2 courses of treatment to assess blood perfusion.

After completion of study treatment, patients are followed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of Solid Tumor or Lymphoma that is metastatic or unresectable; if assessing a single target lesion, histological confirmation of that particular lesion MUST be carried out
* Patients may have received an unlimited number of prior therapies; however, At least 4 weeks MUST have passed since the last chemotherapy to day 1 of registration (6 weeks for regimens containing nitrosoureas or Mitomycin C)
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2.0 mg/dL (does NOT apply to patients with Gilbert's Syndrome)
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal (Patients with liver involvement will be allowed =< 5.0 X institutional upper normal limit)
* Serum creatinine =< 2.0 mg/dL
* Patients MUST have recovered from all treatment related toxicities to Grade 1 NCI CTC (v 4.0) in severity
* Patients must be willing and able to review, understand, and provide written consent before starting therapy
* Patients with stable brain metastasis (stable disease on one MRI assessment at least 4 weeks after completion of whole brain radiation, no evidence of progression on MRI assessment 4 weeks after stereotactic radiosurgery or complete surgical excision) will also be allowed to participate in this trial
* Patients with histologically proven intracranial glioblastoma, gliosarcoma or anaplastic astrocytoma will be eligible; patients must have shown unequivocal radiographic evidence for tumor progression by MRI scan; scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days; if the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required

Exclusion Criteria:

* Patients with squamous non-small cell lung carcinoma
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days of day 1 of registration
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 registration
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to day 1 of therapy
* Patients may not be receiving any other investigational agents
* Patients with bleeding diathesis (clinical bleeding, prothrombin time >= 1.5 X upper institutional normal value, INR >= 1.5, activated partial thromboplastin time aPTT >= 1.5 X upper institutional normal value), active gastric or duodenal ulcer
* Uncontrolled systemic vascular hypertension (Systolic blood pressure > 140 mmHg, Diastolic Blood Pressure > 90 mmHg)
* Urine protein should be screened by dipstick or urine analysis; for proteinuria > 1+ or urine protein:creatinine ratio > 1.0, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on Day 1
* Patients with clinically significant cardiovascular disease:

  * History of CVA within 6 months
  * Myocardial Infarction or unstable angina within 6 months
  * New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Clinically significant peripheral vascular disease
  * QTc prolongation > 500msec or other significant ECG abnormality noted within 14 days of registration
  * Conditions requiring concurrent use of drugs or biologics with proarrythmic potential; these drugs are prohibited during studies with AZD2171 (refer to appendix V for a listing of these agents)
* Patients with history of hemoptysis
* Patients with tumor mass abutting a major vessel
* Pregnant women are excluded from this study because AZD-2171 is an angiogenesis inhibiting agent with potential teratogenic or abortifacient effects; because of the potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD-2171, breastfeeding should be discontinued if the mother is treated with AZD-2171; these potential risks may also apply to other agents used in this study; women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-05; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity profile of combination bevacizumab and cediranib maleate | Up to 6 weeks post-treatment
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Pharmacokinetic profile of oral cediranib maleate in combination with bevacizumab | Baseline and at 1, 2, 3, 4, 6, 8, and 24 hours after cediranib maleate treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States